CLINICAL TRIAL: NCT00333099
Title: Effect of Enteral Immunonutrition During Chemoradiotherapy in Patients With Head and Neck Cancer or Esophageal Cancer
Brief Title: INEC Study: Immuno-modulating Enteral Nutrition in Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fonds National d'Aménagement et de Développement du territoire (FNADT) (Unknown); European Regional Development Fund (Other); Centre Jean Perrin (Other); Centre Leon Berard (Other); Institut de Cancérologie de la Loire (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Hôpital Edouard Herriot (Other); University Hospital, Grenoble (Other); Orkyn' (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHU63-0012
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Malnutrition; Esophageal Cancer; Head and Neck Cancer
Keywords: Enteral nutrition; immunonutrients; head and neck cancer; esophageal cancer; chemoradiotherapy; H&N or esophageal cancer patients with a chemoradiotherapy treatment.
MeSH Terms: conditions — Malnutrition; Esophageal Neoplasms; Head and Neck Neoplasms | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- nutrition (Placebo Comparator): study of immuno-modulating enteral nutrition
  Interventions: Dietary Supplement: Impact (R) Enteral Nutrition; Other: impact

INTERVENTIONS:
Dietary Supplement: Impact (R) Enteral Nutrition — mucositis frequency, treatment tolerance
Other: impact — 1500 calories every day :
  -5 days before the begining of the chemoradiotherapy and until the last day of the treatment

SUMMARY:
The aim of this study is to investigate if enteral immunonutrition of head and neck or esophageal cancer patients, using an arginine, omega 3 fatty acid, nucleotides-enhanced diet [Impact (R), Novartis] versus a standard enteral nutrition (control, Novartis), could improve clinical outcomes (mucositis frequency, treatment tolerance), nutritional and immune status, and life quality parameters.

DETAILED DESCRIPTION:
Malnutrition is frequent in head and neck (H&N) and esophageal cancers and alters immune status, anti-infectious and anti-tumoral defenses and the response to the treatment (surgery, chemotherapy, radiotherapy). Treatment of these 2 types of cancer is often chemoradiotherapy which frequently induces mucositis. Mucositis enhances nutritional risk and could impose a modification or an interruption of the treatment. The aim of this study is to investigate if enteral immunonutrition of head and neck or esophageal cancer patients, using an arginine, omega 3 fatty acid, nucleotides-enhanced diet [Impact(R), Novartis] versus a standard enteral nutrition (control, Novartis), could improve clinical outcomes (mucositis frequency, treatment tolerance), nutritional and immune status, and life quality parameters.

ELIGIBILITY:
Inclusion Criteria:

* H&N and esophageal cancer patients, not treated by surgery and needing chemoradiotherapy
* Performance status: Objective Mucositis Score (OMS) of 0, 1, 2 or Karnofsky > 50%
* Acceptance of a gastrostomy, jejunostomy or a nasogastric tube to conduct enteral nutrition
* Informed consent form signed

Exclusion Criteria:

* H&N cancer treated by exclusive radiotherapy
* H&N and esophageal cancer which can be treated by exclusive surgery
* Tonsil cancer
* Existence of metastases
* Concomitant cancer
* Repeat of cancer at site
* Insulin dependant diabetes
* Thyroid diseases
* Subjects with major surgery or severe infectious status in the 3 preceding months
* Biological assessment incompatible with the esophagus chemotherapy treatment (polynuclear cells < 1500/ml; blood platelets < 100000/ml; serum creatinine > 130 µmol/ml; ASAT, ALAT, ALP and bilirubin > twice the norm)
* Patients taking food or supplements enriched with omega 3 (arginine and nucleotides), during the period of the study and in the preceding month
* Breast feeding women or in period of fertility without effective means of contraception
* Patients who refuse to participate or are unable to receive information or are unable to sign written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-05; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Frequency and grade of mucositis | each visit

SECONDARY OUTCOMES:
Effect on treatment conditions (interruption, doses) | each visit
Other complications linked to chemoradiotherapy | each week of chemoradiotherapy
Nutritional and immune status | at randomisation's visit, visit at the end of treatment, 1, 6 and 12 months after the end of treatment
Life quality | at randomisation's visit, visit at the end of treatment, 6 and 12 months after the end of treatment
Cost | each visit

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Bouteloup, Doctor, Principal Investigator — Hotel Dieu Service d'Hepato-Gastro-Enterologie (service du Pr G. Bommelaer) Clermont-Ferrand; Marie-Paule Vasson, Professor, Study Director — CLAN, Unité de Nutrition, Centre Jean Perrin (Clermont-Ferrand)
Locations (1):
- Hotel Dieu, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] van Bokhorst-de van der Schuer, van Leeuwen PA, Kuik DJ, Klop WM, Sauerwein HP, Snow GB, Quak JJ. The impact of nutritional status on the prognoses of patients with advanced head and neck cancer. Cancer. 1999 Aug 1;86(3):519-27. PMID 10430262
- [Background] Nozoe T, Kimura Y, Ishida M, Saeki H, Korenaga D, Sugimachi K. Correlation of pre-operative nutritional condition with post-operative complications in surgical treatment for oesophageal carcinoma. Eur J Surg Oncol. 2002 Jun;28(4):396-400. doi: 10.1053/ejso.2002.1257. PMID 12099649
- [Background] Gianotti L, Braga M, Nespoli L, Radaelli G, Beneduce A, Di Carlo V. A randomized controlled trial of preoperative oral supplementation with a specialized diet in patients with gastrointestinal cancer. Gastroenterology. 2002 Jun;122(7):1763-70. doi: 10.1053/gast.2002.33587. PMID 12055582
- [Background] de Luis DA, Arranz M, Aller R, Izaola O, Cuellar L, Terroba MC. Immunoenhanced enteral nutrition, effect on inflammatory markers in head and neck cancer patients. Eur J Clin Nutr. 2005 Jan;59(1):145-7. doi: 10.1038/sj.ejcn.1602034. PMID 15266308
- [Derived] Talvas J, Garrait G, Goncalves-Mendes N, Rouanet J, Vergnaud-Gauduchon J, Kwiatkowski F, Bachmann P, Bouteloup C, Bienvenu J, Vasson MP. Immunonutrition stimulates immune functions and antioxidant defense capacities of leukocytes in radiochemotherapy-treated head & neck and esophageal cancer patients: A double-blind randomized clinical trial. Clin Nutr. 2015 Oct;34(5):810-7. doi: 10.1016/j.clnu.2014.12.002. Epub 2014 Dec 9. PMID 25575640
- [Derived] Vasson MP, Talvas J, Perche O, Dillies AF, Bachmann P, Pezet D, Achim AC, Pommier P, Racadot S, Weber A, Ramdani M, Kwiatkowski F, Bouteloup C. Immunonutrition improves functional capacities in head and neck and esophageal cancer patients undergoing radiochemotherapy: a randomized clinical trial. Clin Nutr. 2014 Apr;33(2):204-10. doi: 10.1016/j.clnu.2013.06.008. Epub 2013 Jun 20. PMID 23849811
- See also: Related Info — http://www.canceropole-clara.com